CLINICAL TRIAL: NCT00440349
Title: A Randomised Trial of Prednisone and Tamoxifen in Patients With Idiopathic Retroperitoneal Fibrosis
Brief Title: Prednisone Versus Tamoxifen in Idiopathic Retroperitoneal Fibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Parma (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR09
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Retroperitoneal Fibrosis
Keywords: Retroperitoneal fibrosis; Tamoxifen; Corticosteroids; Obstructive uropathy; Periaortic fibrosis; Chronic periaortitis
MeSH Terms: conditions — Retroperitoneal Fibrosis | interventions — Tamoxifen; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tamoxifen
Drug: Prednisone

SUMMARY:
Idiopathic retroperitoneal fibrosis (IRF) is a rare disease characterised by the presence of a retroperitoneal periaortic fibro-inflammatory tissue which may entrap the ureters and cause renal failure. The treatment of IRF is not well established. Corticosteroids are frequently used, but the anti-estrogen agent tamoxifen has also been reported to be effective in a number of reports. However, no randomised trials have been published so far. The aim of the present study is to compare the efficacy of prednisone and tamoxifen in the treatment of IRF.

DETAILED DESCRIPTION:
Idiopathic retroperitoneal fibrosis (IRF) is a rare condition hallmarked by the presence of a retroperitoneal mass consisting of chronic inflammatory infiltrate and abundant fibrous tissue. IRF usually presents as a systemic inflammatory disease, with constitutional symptoms (e.g. fatigue, weight loss) and high acute-phase reactants; in addition, IRF patients often complain of abdominal or lumbar pain and, if ureteral involvement is present, they may also show oliguria and symptoms related to uremia.

Ureteral obstructive disease is usually managed by placement of ureteral indwelling stents, nephrostomy tubes or, in the more severe cases, surgical ureterolysis. These approaches are usually followed by medical treatment.

The medical treatment of IRF is largely empirical: corticosteroids are routinely used, but a number of reports have shown that tamoxifen may also be effective. However, no prospective controlled trials have been conducted in patients with this condition. In this study, we compare the efficacy of prednisone and tamoxifen in IRF patients.

Patients who received a diagnosis of IRF will be enrolled, while patients with secondary forms of retroperitoneal fibrosis (e.g. drugs, infections, radiotherapy) will be excluded. When present, ureteral obstruction will be managed by ureteral stents/nephrostomy/ureterolysis. All patients will then receive oral prednisone (1 mg/kg/day) for one month, at the end of which they will be randomized to receive either tamoxifen (0.5 mg/kg/day at fixed dose for 8 months) or prednisone (0.5 mg/kg/day for the first month, 0.25 mg/kg/day for the second and third months, and then tapered off during the ensuing 5 months). A CT/MRI study will be performed before the start of treatment, four months after randomization and at the end of treatment. All patients will be followed up for at least 18 months after the end of treatment.

Disease remission will be defined on the basis of clinical symptoms related to IRF (e.g. pain, constitutional symptoms), levels of acute-phase reactants (erythrocyte sedimentation rate, C-reactive protein), and ureteral obstruction (as assessed by sonography or CT/MRI scan).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic or perianeurismal retroperitoneal fibrosis

Exclusion Criteria:

* Previously treated patients; retroperitoneal fibrosis secondary to drugs(e.g. methysergide, methyldopa, pergolide, ergot alkaloids), infections (e.g. tuberculosis), cancer (e.g. lymphoma, sarcoma), radiotherapy, trauma, major surgery, systemic connective tissue or vasculitis disease (e.g. SLE, panarteritis nodosa); pregnancy; active infections or tumours; known hypersensitivity to prednisone or tamoxifen; uncontrolled diabetes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38
Dates: Start 2000-10; Study Completion 2007-04

PRIMARY OUTCOMES:
Difference in recurrence rate at the end of treatment

SECONDARY OUTCOMES:
Difference in reduction in size of IRF (as assessed by CT/MRI)
Difference in renal function

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Buzio, MD, Principal Investigator — University of Parma
Locations (1):
- Department of Clinical Medicine Nephrology and Health Science, Parma University Hospital, Parma, Parma, Italy

REFERENCES:
- [Background] van Bommel EF, Hendriksz TR, Huiskes AW, Zeegers AG. Brief communication: tamoxifen therapy for nonmalignant retroperitoneal fibrosis. Ann Intern Med. 2006 Jan 17;144(2):101-6. doi: 10.7326/0003-4819-144-2-200601170-00007. PMID 16418409
- [Background] Vaglio A, Salvarani C, Buzio C. Retroperitoneal fibrosis. Lancet. 2006 Jan 21;367(9506):241-51. doi: 10.1016/S0140-6736(06)68035-5. PMID 16427494
- [Background] Vaglio A, Buzio C. Chronic periaortitis: a spectrum of diseases. Curr Opin Rheumatol. 2005 Jan;17(1):34-40. doi: 10.1097/01.bor.0000145517.83972.40. PMID 15604902
- [Background] Kardar AH, Kattan S, Lindstedt E, Hanash K. Steroid therapy for idiopathic retroperitoneal fibrosis: dose and duration. J Urol. 2002 Aug;168(2):550-5. PMID 12131307
- [Background] Moroni G, Gallelli B, Banfi G, Sandri S, Messa P, Ponticelli C. Long-term outcome of idiopathic retroperitoneal fibrosis treated with surgical and/or medical approaches. Nephrol Dial Transplant. 2006 Sep;21(9):2485-90. doi: 10.1093/ndt/gfl228. Epub 2006 May 15. PMID 16702201
- [Derived] Vaglio A, Palmisano A, Alberici F, Maggiore U, Ferretti S, Cobelli R, Ferrozzi F, Corradi D, Salvarani C, Buzio C. Prednisone versus tamoxifen in patients with idiopathic retroperitoneal fibrosis: an open-label randomised controlled trial. Lancet. 2011 Jul 23;378(9788):338-46. doi: 10.1016/S0140-6736(11)60934-3. Epub 2011 Jul 4. PMID 21733570